CLINICAL TRIAL: NCT00400751
Title: Phase 1 Study of Family Consultation for Change-Resistant Smokers
Brief Title: Family Consultation for Health-Compromised Smokers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Arizona (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R21DA013121 (NIH)
Record Dates: First submitted 2006-11-15; First posted 2006-11-17 (Estimated); Last update posted 2006-11-17 (Estimated); Status verified 1999-09

CONDITIONS: Nicotine Dependence
Keywords: Health-compromised smokers, family cessation intervention
MeSH Terms: conditions — Tobacco Use Disorder

INTERVENTIONS:
Behavioral: FAMCON (Family Consultation)

SUMMARY:
Although spousal support predicts the success of a smoker's cessation efforts, "social support" interventions based on teaching partners better support skills have had consistently disappointing results. We examined the potential utility of a family-consultation (FAMCON) intervention based on family-systems theory in a treatment-development project involving 20 couples in which one partner (the primary smoker) continued to smoke despite having or being at significant risk for heart or lung disease. Results were promising. The 50% rate of stable abstinence achieved by primary smokers over at least 6 months exceeds benchmark success rates reported in the literature for other, comparably intensive interventions, suggesting that a couple-focused intervention different in concept and format from social-support interventions tested in the past may hold promise for health-compromised smokers. The FAMCON approach appeared particularly well-suited to female smokers and smokers whose partner also smoked - two sub-groups at high risk for relapse.

DETAILED DESCRIPTION:
Although spousal support predicts the success of a smoker's cessation efforts, "social support" interventions based on teaching partners better support skills have had consistently disappointing results. In this Stage I (treatment development) study we examined the potential utility of a family-consultation (FAMCON) intervention based on family-systems theory.

Specifically, in this Phase-I study we developed, standardized, and pilot tested a systemic, couple-focused treatment for change-resistant smokers based on the assumption that a smoker's marital and family relationships play a key role in whether he or she continues to smoke.

The intervention provides up to 10 sessions of "family consultation" over 2-5 months to single- or dual-smoker couples in which at least one partner continued to smoke despite having lung disease, heart disease, or multiple cardiac risk factors.

The treatment focuses on the immediate social context of smoking, aiming both to interrupt well-intended "solutions" that ironically feed back to keep smoking going, and to help clients realign important relationships in ways not organized around tobacco use.

Participants were 20 couples in which one partner (the primary smoker) continued to smoke despite having or being at significant risk for heart or lung disease.

Results are promising. The 50% rate of stable abstinence achieved by primary smokers over 6 months (with 63% abstinence rates for secondary smokers) exceeds benchmark success rates reported in the literature for other, comparably intensive interventions, suggesting that a couple-focused intervention different in concept and format from social-support interventions tested in the past may hold promise for health-compromised smokers. The12-month cessation rates were 40% for primary smokers and 63% for secondary smokers.

The FAMCON approach appeared particularly well-suited to female smokers and smokers whose partner also smoked - two sub-groups at high risk for relapse.

References:

Rohrbaugh, M.J., Shoham, V., Trost, S., Muramoto, M., Cate, R., & Leischow, S. (2001). Couple-dynamics of change resistant smoking: Toward a family-consultation model. Family Process, 40, 15 - 31.

Shoham, V., Rohrbaugh, M.J., Trost, S.E., & Muramoto, M. (in press). A family consultation (FAMCON) intervention for health-compromised smokers. Journal of Substance Abuse Treatment.

ELIGIBILITY:
Inclusion Criteria:

* patient has a diagnosed heart/lung problem or 2+ CAD risk factors
* patient smoked at least 10 cigarettes per day on average for the previous 6 months
* couple married or living in a committed relationship for at least 2 years
* both partners at least 30 years old
* both partners able to read and speak English
* both partners willing to participate in FAMCON
* at least one smoker in the couple hopes to quit within the next two years

Exclusion Criteria:

* terminal illness with life expectancy less that 5 years
* pregnancy
* history of mania or psychosis

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 1999-09; Study Completion 2003-05

PRIMARY OUTCOMES:
Point-Prevalence (PP): 30-day abstinence: Smoker and spouse report
Percent days abstinence Smoker and spouse report
Urges to smoke (self reports)

SECONDARY OUTCOMES:
Health (SF-36)
Marital Satisfaction (Hendrick & Hendrick, 1993)
State Relationship Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Varda Shoham, Ph.D., Principal Investigator — University of Arizona; Michael J. Rohrbaugh, Ph.D., Study Director — University of Arizona
Locations (1):
- University of Arizona, Family Research Laboratory, Dept of Psychology, Tucson, Arizona, United States